CLINICAL TRIAL: NCT06960642
Title: Early Rehabilitation of Intensive Care Unit Patients - a Multinational Prospective Observational Study on Dosage and Outcome
Brief Title: Dosage of Early Rehabilitation of ICU Patients
Acronym: ERUPT
Status: Not yet recruiting | Type: Observational
Sponsor: Medical University of Vienna (Other)
Collaborators: European Society of Intensive Care Medicine (Other)
Responsible Party: Principal Investigator, Stefan Schaller, Professor of Anaesthesia and Anaesthesiological Intensive Care Medicine, Medical University of Vienna
Other Study IDs: ERUPT
Record Dates: First submitted 2025-03-20; First posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Critical Care, Intensive Care; Critical Illness; Physiotherapy; Early Ambulation; Interprofessional Team Collaboration
Keywords: early ambulation; early rehabilitation; early mobilisation; physiotherapy; Physical Therapy; ICUAW; PICS; Intensive Care Unit Acquired Weakness; Post Intensive Care Syndrom; Physical Function; Critical Care; Interprofessional; Nursing
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Independent: Patients who have been functionally independent before ICU admission
- Dependent: Patients who have been functionally dependent before ICU admissoin

SUMMARY:
Rehabilitation already begins in the intensive care unit (ICU) to maintain or restore the functional capacity of ICU patients and to counteract the long-term effects of intensive care treatment. Mobilisation is an important component.

The aim of this multinational observational study is to record and evaluate the different mobilisation practices for ICU patients worldwide. The investigators want to find out which forms of mobilisation in intensive care patients achieve the best results in terms of physical function, functional status and quality of life.

The goal is to recruit over 6,000 patients internationally. No interventions will be carried out, only routine clinical data will be documented and standardised and already established physical tests and questionnaires will be used.

DETAILED DESCRIPTION:
Intensive care treatment can have long-term effects on patients. Around 40% of intensive care unit (ICU) patients develop an Intensive Care Unit Acquired Weakness (ICUAW), which leads to functional limitations and an impairment of independence, participation in everyday life, quality of life and ability to work. Recent studies have shown that early mobilisation has a positive effect on the course of the disease, including improved physical function and independence, shorter ventilation times, and shorter ICU and hospital stays. However, there is currently no standardised approach to mobilisation and the dosage required to achieve the best health outcomes in ICU patients is unknown. There is also a lack of data on patients who were functionally dependent before hospital admission and on patients who were not on invasive mechanical ventilation.

The main objectives of the observational study are:

1. Assessment of the variety of different mobilisation practices worldwide.
2. The analysis of the association of mobilisation dosage on patient outcomes.
3. The evaluation of the association of the prehospital functional status or invasive mechanical ventilation on patient outcomes.

The investigators aim to recruit over 6,000 patients internationally from a minimum of 200 intensive care units. The total duration of the study is 21 months, with participation per patients being 90 days. Routine clinical data and mobilisation data from ICU will be documented, and standardised functional tests and questionnaires will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥ 18 years old) within 48 hours of ICU admission
* Expected to stay > 24 hours in the ICU

Exclusion Criteria:

* Patients who receive end-of-life care at the time of screening
* Patients whose treatment plans are still under discussion and/or not all team members are committed to full active treatment
* Patients whose functional status is unlikely to be obtainable
* Patients with language barriers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intensive care unit patients
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Physical function at ICU discharge | ICU discharge (up to Day 28)
  Physical function measured with the Functional Status Score for the Intensive Care Unit (FSS-ICU). The total score ranges from 0 to 35, with higher scores indicating better physical function.

SECONDARY OUTCOMES:
Highest level of mobility at ICU discharge and 90 days | ICU discharge (up to Day 28) and Day 90
  Highest level of mobility measured with the ICU Mobility Scale (IMS). The scale ranges from 0 to 10, with higher scores indicating a higher level of mobility (up to independent walking).
Physical function at 90 days | Day 90
  Physical function measured with the Functional Status Score for the Intensive Care Unit (FSS-ICU). The total score ranges from 0 to 35, with higher scores indicating better physical function.
Frailty/ Functional status at ICU discharge and 90 days | ICU discharge (up to Day 28) and Day 90
  Frailty/ Functional status measured with the Clinical Frailty Scale (CFS). The scale ranges from 1 (very fit) to 9 (terminally ill), with higher scores indicating a higher degree of frailty.
ICU LOS | ICU admission until ICU discharge (up to Day 28)
  Length of stay in the ICU
Hospital LOS | ICU admission until hospital discharge
  Length of stay in the hospital
ICU mortality | ICU admission until ICU discharge (up to Day 28)
  Mortality during ICU stay
Hospital mortality | ICU admission until hospital discharge
  Mortality during hospital stay
90-day mortality | Day 90
  Mortality at day 90
Disability at 90 days | Day 90
  Disability measured with the WHO Disability Assessment Schedule 2.0 (WHODAS 2.0, 12-item version). Each item is rated on a scale from 1 (no difficulty) to 5 (extreme or cannot do), with higher scores indicating greater disability.
Activities of Daily Living (ADLs) at ICU discharge and 90 days | ICU discharge (up to Day 28) and Day 90
  Activities of Daily Living (ADLs) measured with the Barthel Score. The total score ranges from 0 to 100, with higher scores indicating less assistance and greater independence in performing ADLs.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan J Schaller, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided
Priority will have requests from within the study group. Other requests for research purposes will be reviewed and have to sign contract including data protection.

REFERENCES:
- See also: Study Webpage English — https://www.erupt-study.eu
- See also: Study Webpage German — https://www.erupt.at